CLINICAL TRIAL: NCT00787826
Title: A Longitudinal Phase 2 Study for the Continued Evaluation of the Safety and Immunogenicity of a Live Francisella Tularensis Vaccine, NDBR 101, Lot 4 in Healthy Adults At-Risk for Exposure to Francisella Tularensis
Brief Title: Continued Safety and Immunogenicity Study of a Live Francisella Tularensis Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-15207.a; FY 07-15 (Other: SIP)
Record Dates: First submitted 2008-11-05; First posted 2008-11-10 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Tularemia
Keywords: Live Vaccine Strain (LVS)
MeSH Terms: conditions — Tularemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccination (Experimental): Live Francisella Tularensis Vaccine
  Interventions: Biological: Live Francisella Tularensis Vaccine

INTERVENTIONS:
Biological: Live Francisella Tularensis Vaccine — Approximately 0.0025 mL of vaccine will be administered percutaneously with a bifurcated needle using 15 pricks on the volar surface of the forearm. Vaccination may be repeated up to two times within the year if successful vaccination is not demonstrated by a positive "take" reaction and a MA titer of ≥ 1:20.
  Other Names: LVS Vaccine

SUMMARY:
This study is designed to determine the safety and immunogenicity of a Live Francisella tularensis Vaccine

DETAILED DESCRIPTION:
Study Objectives:

1. To assess the safety of live F. tularensis vaccine NDBR 101.
2. To assess the immunogenicity of live F. tularensis vaccine NDBR 101.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Females of childbearing potential must agree to have a urine or serum pregnancy test on vaccination day, immediately before vaccination (Exception: documented hysterectomy or > 3 years of menopause). The results must be negative. Subjects must agree not to become pregnant for 3 months after receipt of the vaccine.
3. Subjects must be at risk for exposure to F. tularensis.
4. Subjects must have an up-to-date (within 1 year) medical history including concomitant medications, physical examination, and laboratory tests on their charts and be medically cleared for participation by an investigator.
5. Subject must be willing to return for all follow-up visits on days 1 and 2, between days 5-9, 12-16, 28-35, and 56-84 (if needed), all visits for serology, and the closeout interview 6 months (±14 days) after vaccination or revaccination.
6. Subject must agree to report any adverse event which may or may not be associated with administration of the test article for at least 28 days after vaccination.

Exclusion Criteria:

1. Over the age of 65 Years.
2. Vaccinated against tularemia within the last 10 years or had a documented, confirmed tularemia infection.
3. Clinically significant abnormal lab results including evidence of hepatitis C, hepatitis B carrier state, or elevated liver function tests (two times the normal range or at the discretion of the PI).
4. Personal history of an immunodeficiency or current treatment with an oral or intravenous immunosuppressive medication.
5. Confirmed HIV* infection.
6. A medical condition that, in the judgment of the Principal Investigator (PI), would impact subject safety.
7. Antibiotic therapy within 7 days before vaccination.
8. Pregnancy or lactation. Subjects must agree not to become pregnant for 3 months after receipt of the vaccine.
9. Any known allergies to any component of the vaccine:

   Modified casein partial hydrolysate medium Glucose cysteine hemin agar Sucrose gelatin agar stabilizer
10. Administration of another vaccine within 4 weeks of tularemia vaccination.
11. Any unresolved AE resulting from a previous immunization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-08-28 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number for adverse events. | 5 years
  The nature (body system affected, type (local or systemic), severity, frequency of occurrence, relationship to vaccine, treatment or intervention offered if any, and resolution or outcome) and frequency of adverse events for the assessment population (all subjects receiving one or more vaccinations under this protocol).
Number of erythematous papule, vesicle, and/or eschar with or without underlying induration | 7 (± 2 days) after vaccination
  Incidence of positive "take" reaction (development of an erythematous papule, vesicle, and/or eschar with or without underlying induration) following vaccination for all subjects regardless of compliance.
Microagglutination (MA) titer that shows a ≥ 4-fold rise in antibody titer after vaccination. | 28-35 days
  Seroconversion will be evaluated for subjects who are compliant with the titer schedule.
  Seroconversion is defined as microagglutination (MA) titer that shows a ≥ 4-fold rise in antibody titer after vaccination.

SECONDARY OUTCOMES:
Number of tularemia cases following exposure to F. tularensis in a successfully vaccinated individual | 5 years
  Documented occurrence of tularemia following exposure to F. tularensis in a successfully vaccinated individual (positive "take" reaction and seroconversion [≥ 4-fold rise in antibody titer after vaccination]).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Cardile, DO, Principal Investigator — USAMRIID Medical Division
Locations (1):
- U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States